CLINICAL TRIAL: NCT04984499
Title: In Vivo Clinical Investigation of the Safety and Performance of Dental Implants TBR® Tissue Level Z1 With Ceramic Emergence
Brief Title: In Vivo Clinical Investigation of the Safety and Performance of Dental Implants TBR® Tissue Level Z1
Acronym: Z1
Status: Active, not recruiting | Type: Observational
Sponsor: Sudimplant SAS - Groupe TBR (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A01926-51
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Edentulous Mouth
MeSH Terms: conditions — Mouth, Edentulous | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dental implant — The procedure used to accomplish its intended use is as follows :
  The recipient implant site is prepared using a drilling sequence, then the implant is placed at the crestal level with a cover screw to allow the tissues healing. After this healing phase, the final prosthesis will be loaded on the implant.

SUMMARY:
Partial or total edentulousness has a significant impact on quality of life both functionally and aesthetically.

TBR® Tissue Level Z1 Implants allow the patient to prevent bone resorption and maintain facial tissue and musculature support. At the functional level, the patient who benefits from implant treatment regains normal masticatory function with all the benefits on the quality of life that this can bring him.

Due to the osseointegration of the implant and the biocompatibility of the materials used, the implant treatment remains effective in the long term and makes it possible to maintain the aesthetics of the smile.

DETAILED DESCRIPTION:
Many adults have one or more missing teeth. The negative consequences of partial or total edentulousness are numerous in the orofacial sphere:

* Edentulousness causes a strong aesthetic deficit due to the lack of support of facial tissues and musculature;
* Edentulousness generates a functional deficit that can have significant repercussions on the nutritional status of the affected subject;
* Edentulousness is accompanied by bone resorption of the jawbones which is inevitable in the absence of implant treatment;
* In addition, the resulting feelings of discomfort and fragility are experienced as a real psychological handicap by the patient, partially or totally edentulous, which can then have significant repercussions on his social life.

TBR® Tissue Level Z1 implants are intended for placement in the maxillary or mandibular arch in partially or completely edentulous patients for prosthetic restoration in the following cases:

* Single edentulousness,
* Intercalary edentulousness,
* Terminal edentulousness,
* Total edentulousness.

The following clinical conditions must be observed before placing a dental implant:

* Sufficient quality and volume of bone support;
* Healthy oral condition;
* no contraindications for implant setting

The procedure used to accomplish its intended use is as follows:

* The receiving implant site is prepared using an established drilling sequence then the implant is placed in this site: the body of the implant (in titanium) has an endosseous position while the ring (in ceramic) remains transgingival;
* After an osseointegration time, the final prosthetic abutment will be loaded on the implant.

The expected benefits of this surgery are to improve the quality of life of patients, to recover the chewing function and the aesthetics of the smile.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient who has completed bone growth
* Patient informed and willing to participate in the study
* Partially or totally toothless patient who will be implanted with the TBR® Bone Level implant(s) for the prospective cohort
* Patient implanted with the TBR® TISSUE LEVEL Z1 implant(s) before June 2011 for the retrospective cohort

Exclusion Criteria:

* Pregnant or lactating women
* Patient with bone disease of the head and neck region
* Patient refusing to participate in the study
* Patient with at least one contraindication to implantation
* Patient on osteoporosis treatment with Biphosphonates or Denosumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient partially or totally toothless
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
the success rate of tissue integration of the implant | 15 years after implantation
  Integration of the implant 15 years after implantation

SECONDARY OUTCOMES:
Change of the quality of life of patients following the recovery of a complete dentition with the OHIP- 14 score (Oral Health Impact Profile) | 5 years after implantation
  The quality of life of patients will be evaluate with the OHIP- 14 score (Oral Health Impact Profile) before implantation and 5 years after implantation
Complication rate taking into account pain, local tenderness, infection, allergy, mobility of the implant, fracture | 5 years after implantation
  pain, local tenderness, infection, allergy, mobility of the implant, fracture will be collected during during the 5 years follow-up
Measuring chewing function with occlusal assessment | 5 years after implantation
  Occlusal assessment will be performed after implantation and at 5 years follow-up
Radiographic analysis of the osseointegration of the implant | 5 years after implantation
  A radiographic analysiswill be performed after implantation and at 5 years follow-up to evaluate the osseointegration of the implant
Absence of inflammation (visual) and infection (radiographic) | 5 years after implantation
  Assessment of inflammation with visual examination and assessment of infection with radiographic examination 5 years after implantation

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet du Dr ALLOUCHE, Montpellier, France